CLINICAL TRIAL: NCT05041855
Title: Family Inclusive Childhood Obesity Treatment Designed for Low Income and Hispanic Families
Brief Title: Childhood Obesity Treatment Designed for Low Income and Hispanic Families
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Colorado State University (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-3721; 1R01DK130176-01 (NIH)
Record Dates: First submitted 2021-09-03; First posted 2021-09-13 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Pediatric Obesity; Healthy Eating; Physical Activity; Minority Health; Mindfulness; Family; Counseling
Keywords: Childhood Obesity; Childhood obesity treatment; Adolescent obesity; Childhood Obesity Prevention; Family; Community; Physical activity; Nutrition; Hispanic; Latino; Motivational Interviewing; Food Insecurity
MeSH Terms: conditions — Pediatric Obesity; Motor Activity | interventions — Primary Health Care

STUDY DESIGN:
Intervention Model Description: Family participants (children and their caregivers) will be randomized to the Healthy Living Program group intervention or the Recommended Treatment of Obesity in Primary Care individual intervention for an observation period of 18 months from baseline.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Community based childhood obesity intervention (Experimental): A novel family-inclusive childhood obesity treatment program consisting of 12 family group sessions delivered in English and Spanish by health educators at community recreation centers, followed by three group booster sessions occurring every 6 months.
  Interventions: Behavioral: The Healthy Living Program/La Vida Saludable
- Primary care based childhood obesity intervention (Active Comparator): A healthy lifestyle counseling intervention delivered by trained primary care providers and health educators at visits occurring every 3 months.
  Interventions: Behavioral: Recommended Treatment of Obesity in Primary Care

INTERVENTIONS:
Behavioral: The Healthy Living Program/La Vida Saludable — A whole-family group childhood obesity intervention delivered at community recreation centers
  Other Names: HeLP
  Arms: Community based childhood obesity intervention
Behavioral: Recommended Treatment of Obesity in Primary Care — A healthy lifestyle counseling protocol that enhances usual primary care
  Other Names: RTOP
  Arms: Primary care based childhood obesity intervention

SUMMARY:
This study is a type-1 hybrid effectiveness-implementation RCT comparing a novel family-inclusive childhood obesity treatment program, the "Healthy Living Program" (HeLP), to a protocol that enhances usual primary care to deliver Recommended Treatment of Obesity in Primary Care (RTOP). Children with obesity and their families will be referred to the study by primary care providers and randomized to HeLP or RTOP. The clinical setting is a practice-based research network serving majority Hispanic and Medicaid-insured populations. The intensive phase and booster sessions of HeLP will take place at recreation centers located near the clinics and will be led by health educators employed by the clinics. Visits with primary care providers (PCPs) for HeLP maintenance or RTOP will occur at the clinics.

DETAILED DESCRIPTION:
This study is a Randomized Controlled Trial (RCT) to learn about how well a family childhood weight management program works compared to healthy lifestyle counseling by providers at participating clinics. The goal is to compare weight change in children with obesity from low-income predominantly Hispanic/Latino families that will participate in the program, the Healthy Living Program (HeLP) vs. Recommended Treatment of Obesity in Primary Care (RTOP). Low-income children with obesity from mostly Hispanic clinical populations will be referred to the project by their primary doctors and will be enrolled into either HeLP or RTOP. Families (including siblings and caregivers) who are in HeLP will be offered 12 sessions at local rec centers where health educators and fitness trainers will teach them about parenting skills, nutrition, fitness, and mindfulness. Families who are in RTOP will receive an enhanced version of the care that is usually provided at their primary care clinics. Providers will be trained in a skill called Motivational Interviewing and use an electronic tool called "HeartSmartKids" to help families make healthy lifestyle changes. Families who are in RTOP will go to follow-up visits every 3 months and will go to HeLP after 18 months.

Aim 1 (Treatment): To compare the BMI change relative to the 95th percentile for age and sex in children with obesity in 3 different age groups (2-6, 7-12, and 13-16 years old) 18 months after being in either HeLP or RTOP.

Aim 2 (Prevention): To compare the weight change in healthy and unhealthy weight 2-6-year-old children who have siblings with obesity and are in either HeLP or RTOP.

Aim 3 (Implementation): To describe implementation processes of HeLP and RTOP using a framework called RE-AIM: R-Reach: Is the project reaching the people it needs to reach? E-Effectiveness: Is the program effective? A-Adoption: are the health educators, providers, and clinics promoting and doing the program? I-Implementation: Are the health educators, providers and clinics delivering the intervention as intended? M-Maintenance: Is the intervention working to help children with their weight and healthy lifestyle changes? The cost of delivering the program will also be studied to inform potential sustainability.

ELIGIBILITY:
Inclusion Criteria:

* Child aged 2-16yrs

  * With overweight or obesity (BMI >85th percentile)
  * Referred by PCP
* Primary Adult Caregiver
* Up to two siblings of any BMI status (if multiple siblings are available, enrollment goals stratified by age and BMI will be used to select siblings for enrollment.)

Exclusion Criteria:

* Parent without fluency in either Spanish or English
* Current participation in a clinically referred obesity treatment program
* Child non-ambulatory, non-verbal, or diagnosed with a genetic syndrome associated with obesity.
* Children with severe depression on initial screening (CES-D >/=40 or suicidal ideation) will be excluded and referred to psychiatric treatment and therapy.
* Children who have been diagnosed by PCP at time of initial screening with severe comorbidities of obesity, including:

  * Type 2 diabetes
  * Stage 2 hypertension
  * Severe hyperlipidemia
  * Severe obstructive sleep apnea will be excluded from the study and directed to the only Tertiary Care Childhood Obesity Treatment program in the state of Colorado: Lifestyle Medicine at Children's Hospital Colorado.

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 554 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in Body Mass Index (BMI) %95 in children with obesity (treatment) | From Baseline to Month 18
  Change in BMI%95 as measured in 2-16 yr old children with obesity BMI%95 is the percentage a child's BMI represents of the BMI value at the 95th percentile for age and sex calculated using the Centers for Disease Control (CDC) program for Statistical Analysis System (SAS).
Change in Body Mass Index (BMI) %95 in healthy and overweight children (prevention) | From Baseline to Month 18
  Change in BMI%95 as measured in healthy and overweight 2-11 yr old siblings of the children with obesity. BMI%95 is the percentage a child's BMI represents of the BMI value at the 95th percentile for age and sex calculated using the CDC program for SAS.

SECONDARY OUTCOMES:
Change in Body Mass Index (BMI) %95 in children with obesity (treatment) | From Baseline to Month 12
  Change in BMI%95 as measured in 2-16 yr old children with obesity BMI%95 is the percentage a child's BMI represents of the BMI value at the 95th percentile for age and sex calculated using the CDC program for SAS.
Change in Body Mass Index (BMI) %95 in healthy and overweight children (prevention) | From Baseline to Month 12
  Change in BMI%95 as measured in healthy and overweight 2-11 yr old siblings of the children with obesity. BMI%95 is the percentage a child's BMI represents of the BMI value at the 95th percentile for age and sex calculated using the CDC program for SAS.
Change in nutrition aspects of the home environment as measured by the Comprehensive Home Environment Survey (CHES) | Baseline, Month 18
  The CHES is a validated parent-report instrument that measures aspects of the home environment influencing child diet and physical activity. Possible scores on the nutrition scale range from 0 to 10, with higher scores indicating a better home environment for nutrition.
Change in physical activity and media aspects of the home environment as measured by the Comprehensive Home Environment Survey (CHES) | Baseline, Month 18
  The CHES is a validated parent-report instrument that measures aspects of the home environment influencing physical activity and media. Possible scores are on a scale from 0 to 8 with higher scores indicating a better home environment for physical activity and media.
Change from Baseline in food insecurity at 18 months as measured by the US Department of Agriculture (USDA) Household Food Security Survey scores | Baseline, Month 18
  The USDA Household Food Security Survey is a validated scale that measures food insecurity. Possible scores range from 0 to 18, with higher scores indicating lower food security.
Change from baseline in Hunger at 18 months as measured by the Three-Factor Eating Questionnaire for Children and Adolescents | Baseline, Month 18
  Three-Factor Eating Questionnaire for Children and Adolescents is a validated scale that measures eating attitudes and behaviors in 3 domains: 'Cognitive Restraint of Eating', 'Disinhibition', and 'Hunger'. Possible scores range from 0-14 for 'Hunger' with higher scores indicating worse eating attitudes and behaviors.
Change from baseline in Cognitive Restraint of Eating at 18 months as measured by the Three-Factor Eating Questionnaire for Children and Adolescents | Baseline, Month 18
  Three-Factor Eating Questionnaire for Children and Adolescents is a validated scale that measures eating attitudes and behaviors in 3 domains: 'Cognitive Restraint of Eating', 'Disinhibition', and 'Hunger'. Possible scores range from 0-21 for 'Cognitive Restraint of Eating' with higher scores indicating worse eating attitudes and behaviors.
Change from baseline in Disinhibition at 18 months as measured by the Three-Factor Eating Questionnaire for Children and Adolescents | Baseline, Month 18
  Three-Factor Eating Questionnaire for Children and Adolescents is a validated scale that measures eating attitudes and behaviors in 3 domains: 'Cognitive Restraint of Eating', 'Disinhibition', and 'Hunger'. Possible scores range from 0-16 for 'Disinhibition' with higher scores indicating worse eating attitudes and behaviors.
Change from baseline in physical fitness at 6 months as measured by the Progressive Aerobic Cardiovascular Endurance Run (PACER) Scores | Baseline, Month 6
  The Progressive Aerobic Cardiovascular Endurance Run (PACER) test measures physical fitness by estimating VO2peak. Scores are based on a shuttle-run of 20 meter intervals. The higher the number of intervals completed in the allotted time indicating a better outcome.
Change from baseline in physical fitness at 18 months as measured by the Progressive Aerobic Cardiovascular Endurance Run (PACER) Scores | Baseline, Month 18
  The Progressive Aerobic Cardiovascular Endurance Run (PACER) test measures physical fitness by estimating VO2peak. Scores are based on a shuttle-run of 20 meter intervals. The higher the number of intervals completed in the allotted time indicating a better outcome.
Change from Baseline in Hemoglobin A1c (HbA1c) blood glucose tests at 18 months | Baseline up to Month 18
  HbA1c blood glucose test, routinely measured as part of pediatric well child care for children 10 years and older with obesity, measures the average level of glucose in blood with normal range 4.2% to 5.6%, prediabetes range 5.7% to 6.4%, and ≥6.5% indicating diabetes. Higher numerical values above 5.7 indicate worse blood sugar control. Investigators will compare the mean A1c between the two groups.
Change from Baseline in Alanine Transaminase (ALT) liver enzyme levels tests at 18 months | Baseline up to Month 18
  ALT levels in the blood, routinely measured as part of pediatric well child care for children 10 years and older with obesity, is measured by milligrams per deciliter (mg/dl) with ALT>22mg/dL in females less than 18 years, and ALT >26 mg/dL in males less than 18 years indicating possible non-alcoholic fatty liver disease. Higher levels of ALT above these normal cutoffs may represent worsening liver disease. Investigators will compare the mean ALT between the two groups.
Change from Baseline in Low Density Lipoprotein (LDL) Cholesterol tests or fasting lipids tests at 18 months | Baseline up to Month 18
  The LDL blood test, routinely measured as part of pediatric well child care for children 10 years and older with obesity, measures cholesterol with an LDL>110 mg/dL in children indicating a worse outcome such as increased long-term risk of heart disease. Higher levels of LDL above these normal cutoffs may represent higher risk of heart disease. Investigators will compare the mean LDL between the two groups.
Change from Baseline in Caregiver Waist Circumference (WC) at 12 months | Baseline, Month 12
  Waist Circumference is measured to classify adults aged 20 or older into 3 health risk categories, low health risk, increased health risk, and high health risk. A higher waist circumference indicates a worse outcome.
Change from Baseline in Caregiver Waist Circumference (WC) at 18 months | Baseline, Month 18
  Waist Circumference is measured to classify adults aged 20 or older into 3 health risk categories, low health risk, increased health risk, and high health risk. A higher waist circumference indicates a worse outcome.
Change from Baseline in Adult Caregiver Body Mass Index (BMI) at 12 months | Baseline, Month 12
  Body Mass Index (BMI) is a person's weight in kilograms divided by the square of their height in meters. Scores between 18.5 and 24.9 indicate a healthy weight. A higher BMI indicates a worse outcome.
Change from Baseline in Adult Caregiver Body Mass Index (BMI) at 18 months | Baseline, Month 18
  Body Mass Index (BMI) is a person's weight in kilograms divided by the square of their height in meters. Scores between 18.5 and 24.9 indicate a healthy weight. A higher BMI indicates a worse outcome.
Change from Baseline to 6 months in levels of Familism as measured by the Pan-Hispanic Familism Scale | Baseline, Month 6
  The Pan-Hispanic Familism Scale is a validated scale that measures familism, a value system found within many Hispanic/Latino communities that emphasizes familial honor, respect, and mutual collaboration. Participants respond on a 5-point Likert scale from 1=Strongly disagree to 5=Strongly Agree. Higher Scores indicate a higher degree of adherence to Familism.
Change from Baseline in 18 months in levels of Familism as measured by the Pan-Hispanic Familism Scale | Baseline, Month 18
  The Pan-Hispanic Familism Scale is a validated scale that measures familism, a value system found within many Hispanic/Latino communities that emphasizes familial honor, respect, and mutual collaboration. Participants respond on a 5-point Likert scale from 1=Strongly disagree to 5=Strongly Agree. Higher Scores indicate a higher degree of adherence to Familism.
Change from Baseline in weight-related quality of life at 6 months as measured by the Sizing Me Up child report | Baseline, Month 6
  Sizing Me Up is a validated weight-related quality of life questionnaire for children aged 10 years and older. Possible scores range from 0 to 100 with higher scores indicating a better quality of life.
Change from Baseline in weight-related quality of life at 18 months as measured by the Sizing Me Up child report | Baseline, Month 18
  Sizing Me Up is a validated weight-related quality of life questionnaire for children aged 10 years and older. Possible scores range from 0 to 100 with higher scores indicating a better quality of life.
Change from Baseline in weight-related quality of life at 6 months as measured by the Sizing Them Up Parent report | Baseline, Month 6
  Sizing Them Up is a validated weight-related quality of life questionnaire for parents/primary caregivers of children 6 to 10 years of age. Possible scores range from 0 to 100 with higher scores indicating a better quality of life.
Change from Baseline in weight-related quality of life at 18 months as measured by the Sizing Them Up Parent report | Baseline, Month 18
  Sizing Them Up is a validated weight-related quality of life questionnaire for parents/primary caregivers of children 6 to 10 years of age. Possible scores range from 0 to 100 with higher scores indicating a better quality of life.
Change from Baseline in depressive symptoms in parents at 6 months as measured by the Center of Epidemiological Studies Depression Scale (CES-D) | Baseline, Month 6
  The Center of Epidemiological Studies Depression Scale is a validated questionnaire that assesses depressive symptoms in parents. Possible scores range from 0-60 with higher scores indicating worse depressive symptoms.
Change from Baseline in depressive symptoms in parents at 18 months as measured by the Center of Epidemiological Studies Depression Scale (CES-D) | Baseline, Month 18
  The Center of Epidemiological Studies Depression Scale is a validated questionnaire that assesses depressive symptoms in parents. Possible scores range from 0-60 with higher scores indicating worse depressive symptoms.
Change from Baseline in depressive symptoms in adolescents 12-18 years at 6 months as measured by the Center of Epidemiological Studies Depression Scale (CES-D) | Baseline, Month 6
  The Center of Epidemiological Studies Depression Scale is a validated questionnaire that assesses depressive symptoms in adolescents 12-18 years. Possible scores range from 0-60 with higher scores indicating worse depressive symptoms.
Change from Baseline in depressive symptoms in adolescents 12-18 years at 18 months as measured by the Center of Epidemiological Studies Depression Scale (CES-D) | Baseline, Month 18
  The Center of Epidemiological Studies Depression Scale is a validated questionnaire that assesses depressive symptoms in adolescents 12-18 years. Possible scores range from 0-60 with higher scores indicating worse depressive symptoms.
Change from Baseline in depressive symptoms in children at 6 months as measured by the Center of Epidemiological Studies Depression Scale for Children 6-12 years (CES-DC) | Baseline, Month 6
  The Center of Epidemiological Studies Depression Scale for Children is a validated questionnaire that measures depressive symptoms in 6-12 year old children. Possible scores range from 0-60 with higher scores indicating worse depressive symptoms.
Change from Baseline in depressive symptoms in children at 18 months as measured by the Center of Epidemiological Studies Depression Scale for Children 6-12 years (CES-DC) | Baseline, Month 18
  The Center of Epidemiological Studies Depression Scale for Children is a validated questionnaire that measures depressive symptoms in 6-12 year old children. Possible scores range from 0-60 with higher scores indicating worse depressive symptoms.
Reach as measured by the proportion of eligible children seen for well-child care that are randomized. | up to Month 18
  Reach as measured by the proportion of children seen for a well-child check at each clinic that are randomized during the study.
Adoption as measured by the proportion of training sessions attended by medical providers | up to month 48
  Number of training sessions that Primary Care Providers attend. Attendance will be taken at all PCP trainings. There will be 4 training sessions within the first 12 months and 2 refresher training sessions between 36-48 months. Total 6 possible sessions attended, with higher attendance rates indicating a better outcome.
Primary Care Visit Frequency in the as measured by number of clinic visits for each child | up to month 36
  Primary Care Visit Frequency, as measured by the number of clinic visits for child weight follow-up reported in Clinic Electronic Medical Records (EMR's.
Change in history of Coronavirus Disease 2019 (COVID-19) diagnosis status in a parent participant | Baseline, up to month 18
  Response to questionnaire administered every 6 months throughout the study period to participating parents querying whether they or any of their participating children have tested positive for COVID-19 using a laboratory assay. Participants with no history of COVID-19 diagnosis at baseline who later report positive diagnosis will be defined as new diagnosis of COVID-19 during the study period.
Change in history of COVID-19 diagnosis status in a child participant | Baseline, up to month 18
  Response to questionnaire administered every 6 months throughout the study period to participating parents querying whether any of their participating children have tested positive for COVID-19 using a laboratory assay. Child participants with no history of COVID-19 diagnosis at baseline whose parents later report positive diagnosis for that child will be defined as new diagnosis of COVID-19 during the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew A Haemer, MD MPH, Principal Investigator — University of Colorado, Denver
Locations (2):
- United States (2):
  - University of Colorado Anschutz, Aurora, Colorado
  - Colorado State University-College of Health and Human Sciences, Fort Collins, Colorado

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kirk S, Zeller M, Claytor R, Santangelo M, Khoury PR, Daniels SR. The relationship of health outcomes to improvement in BMI in children and adolescents. Obes Res. 2005 May;13(5):876-82. doi: 10.1038/oby.2005.101. PMID 15919841
- [Background] Stevens VJ, Glasgow RE, Toobert DJ, Karanja N, Smith KS. Randomized trial of a brief dietary intervention to decrease consumption of fat and increase consumption of fruits and vegetables. Am J Health Promot. 2002 Jan-Feb;16(3):129-34. doi: 10.4278/0890-1171-16.3.129. PMID 11802257
- [Background] Fontaine KR, Redden DT, Wang C, Westfall AO, Allison DB. Years of life lost due to obesity. JAMA. 2003 Jan 8;289(2):187-93. doi: 10.1001/jama.289.2.187. PMID 12517229
- [Background] Finkelstein EA, Khavjou OA, Thompson H, Trogdon JG, Pan L, Sherry B, Dietz W. Obesity and severe obesity forecasts through 2030. Am J Prev Med. 2012 Jun;42(6):563-70. doi: 10.1016/j.amepre.2011.10.026. PMID 22608371
- [Background] Gilbert, K., et al., Using Health IT to bridge clinic and community in the fight against childhood obesity, in American Public Health Association. 2012: San Francisco. p. publication #268558.
- [Background] Haemer, M., et al. Controlled Trial of Technology Supported Motivational Interviewing for Childhood Obesity. in The Obesity Society. 2013. Atlanta, GA.
- [Background] Davidson AJ, McCormick EV, Dickinson LM, Haemer MA, Knierim SD, Hambidge SJ. Population-level obesity surveillance: monitoring childhood body mass index z-score in a safety-net system. Acad Pediatr. 2014 Nov-Dec;14(6):632-8. doi: 10.1016/j.acap.2014.06.007. Epub 2014 Oct 30. PMID 25439162
- [Background] Cason-Wilkerson R, Goldberg S, Albright K, Allison M, Haemer M. Factors influencing healthy lifestyle changes: a qualitative look at low-income families engaged in treatment for overweight children. Child Obes. 2015 Apr;11(2):170-6. doi: 10.1089/chi.2014.0147. Epub 2015 Feb 25. PMID 25715107
- [Background] Knierim SD, Rahm AK, Haemer M, Raghunath S, Martin C, Yang A, Clarke C, Hambidge SJ. Latino parents' perceptions of weight terminology used in pediatric weight counseling. Acad Pediatr. 2015 Mar-Apr;15(2):210-7. doi: 10.1016/j.acap.2014.11.003. Epub 2014 Dec 20. PMID 25536907
- [Background] Haemer, M., et al., Beyond 5210: Results of Universal Lifestyle Screening in Community Health Centers, in Pediatric Academic Societies. 2016: Baltimore, MD.
- [Background] Cardel MI, Tong S, Pavela G, Dhurandhar E, Miller D, Boles R, Haemer M. Youth Subjective Social Status (SSS) is Associated with Parent SSS, Income, and Food Insecurity but not Weight Loss Among Low-Income Hispanic Youth. Obesity (Silver Spring). 2018 Dec;26(12):1923-1930. doi: 10.1002/oby.22314. Epub 2018 Nov 13. PMID 30421861
- [Background] Haemer, M., et al., Mixed Methods Study of Motivational Interviewing Training on Providers' Counseling for Healthy Weight, in Pediatric Academic Societies. 2018: Toronto, Ontario.
- [Background] Knierim SD, Newcomer S, Castillo A, Rahm AK, Raghunath S, Clarke C, Wright L, Haemer M, Hambidge SJ. Latino Parents' Perceptions of Pediatric Weight Counseling Terms. Acad Pediatr. 2018 Apr;18(3):342-353. doi: 10.1016/j.acap.2017.09.006. Epub 2017 Sep 12. PMID 28919572
- [Background] Nederveld A, Cox-Martin M, Bayliss E, Allison M, Haemer M. Food Insecurity and Healthy Behavior Counseling in Primary Care. J Health Dispar Res Pract. 2018 Fall;11(3):49-58. PMID 34295574
- [Background] Moore, J., et al., Weight-Related Quality of Life in a Community-Based Weight Management Trial among Underserved Youth, in The Obesity Society. 2019: Las Vegas, NV.
- [Background] Steen, E., et al. Communication Characteristics of Parents of Latino Preschoolers that Predict Improved Readiness to Change for Child Weight After a Clinic Visit. in American Society for Nutrition. 2020. Seattle WA.
- [Background] Curran GM, Bauer M, Mittman B, Pyne JM, Stetler C. Effectiveness-implementation hybrid designs: combining elements of clinical effectiveness and implementation research to enhance public health impact. Med Care. 2012 Mar;50(3):217-26. doi: 10.1097/MLR.0b013e3182408812. PMID 22310560
- [Background] Barlow SE; Expert Committee. Expert committee recommendations regarding the prevention, assessment, and treatment of child and adolescent overweight and obesity: summary report. Pediatrics. 2007 Dec;120 Suppl 4:S164-92. doi: 10.1542/peds.2007-2329C. PMID 18055651
- [Background] Spear BA, Barlow SE, Ervin C, Ludwig DS, Saelens BE, Schetzina KE, Taveras EM. Recommendations for treatment of child and adolescent overweight and obesity. Pediatrics. 2007 Dec;120 Suppl 4:S254-88. doi: 10.1542/peds.2007-2329F. PMID 18055654
- [Background] Glasgow RE, Vogt TM, Boles SM. Evaluating the public health impact of health promotion interventions: the RE-AIM framework. Am J Public Health. 1999 Sep;89(9):1322-7. doi: 10.2105/ajph.89.9.1322. PMID 10474547
- [Background] Glasgow RE, Harden SM, Gaglio B, Rabin B, Smith ML, Porter GC, Ory MG, Estabrooks PA. RE-AIM Planning and Evaluation Framework: Adapting to New Science and Practice With a 20-Year Review. Front Public Health. 2019 Mar 29;7:64. doi: 10.3389/fpubh.2019.00064. eCollection 2019. PMID 30984733
- [Background] Shomaker LB, Pivarunas B, Annameier SK, Gulley L, Quaglia J, Brown KW, Broderick P, Bell C. One-Year Follow-Up of a Randomized Controlled Trial Piloting a Mindfulness-Based Group Intervention for Adolescent Insulin Resistance. Front Psychol. 2019 May 8;10:1040. doi: 10.3389/fpsyg.2019.01040. eCollection 2019. PMID 31133946
- [Background] Pinard CA, Yaroch AL, Hart MH, Serrano EL, McFerren MM, Estabrooks PA. The Validity and reliability of the Comprehensive Home Environment Survey (CHES). Health Promot Pract. 2014 Jan;15(1):109-17. doi: 10.1177/1524839913477863. Epub 2013 Mar 7. PMID 23471699
- [Background] Resnicow K, McMaster F, Woolford S, Slora E, Bocian A, Harris D, Drehmer J, Wasserman R, Schwartz R, Myers E, Foster J, Snetselaar L, Hollinger D, Smith K. Study design and baseline description of the BMI2 trial: reducing paediatric obesity in primary care practices. Pediatr Obes. 2012 Feb;7(1):3-15. doi: 10.1111/j.2047-6310.2011.00001.x. Epub 2011 Dec 13. PMID 22434735
- [Background] Schwartz RP, Hamre R, Dietz WH, Wasserman RC, Slora EJ, Myers EF, Sullivan S, Rockett H, Thoma KA, Dumitru G, Resnicow KA. Office-based motivational interviewing to prevent childhood obesity: a feasibility study. Arch Pediatr Adolesc Med. 2007 May;161(5):495-501. doi: 10.1001/archpedi.161.5.495. PMID 17485627
- [Background] Resnicow K, Harris D, Wasserman R, Schwartz RP, Perez-Rosas V, Mihalcea R, Snetselaar L. Advances in Motivational Interviewing for Pediatric Obesity: Results of the Brief Motivational Interviewing to Reduce Body Mass Index Trial and Future Directions. Pediatr Clin North Am. 2016 Jun;63(3):539-62. doi: 10.1016/j.pcl.2016.02.008. PMID 27261549
- [Background] Resnicow K, McMaster F, Bocian A, Harris D, Zhou Y, Snetselaar L, Schwartz R, Myers E, Gotlieb J, Foster J, Hollinger D, Smith K, Woolford S, Mueller D, Wasserman RC. Motivational interviewing and dietary counseling for obesity in primary care: an RCT. Pediatrics. 2015 Apr;135(4):649-57. doi: 10.1542/peds.2014-1880. PMID 25825539
- [Background] Klein JD, Sesselberg TS, Johnson MS, O'Connor KG, Cook S, Coon M, Homer C, Krebs N, Washington R. Adoption of body mass index guidelines for screening and counseling in pediatric practice. Pediatrics. 2010 Feb;125(2):265-72. doi: 10.1542/peds.2008-2985. Epub 2010 Jan 18. PMID 20083518
- [Background] Runkle C, Osterholm A, Hoban R, McAdam E, Tull R. Brief negotiation program for promoting behavior change: the Kaiser Permanente approach to continuing professional development. Educ Health (Abingdon). 2000;13(3):377-86. doi: 10.1080/135762800750059499. PMID 14742064
- [Background] Lozano P, McPhillips HA, Hartzler B, Robertson AS, Runkle C, Scholz KA, Stout JW, Kieckhefer GM. Randomized trial of teaching brief motivational interviewing to pediatric trainees to promote healthy behaviors in families. Arch Pediatr Adolesc Med. 2010 Jun;164(6):561-6. doi: 10.1001/archpediatrics.2010.86. PMID 20530307
- [Background] Arora S, Kalishman SG, Thornton KA, Komaromy MS, Katzman JG, Struminger BB, Rayburn WF, Bradford AM. Project ECHO: A Telementoring Network Model for Continuing Professional Development. J Contin Educ Health Prof. 2017 Fall;37(4):239-244. doi: 10.1097/CEH.0000000000000172. PMID 29189491
- [Background] Freedman DS, Butte NF, Taveras EM, Lundeen EA, Blanck HM, Goodman AB, Ogden CL. BMI z-Scores are a poor indicator of adiposity among 2- to 19-year-olds with very high BMIs, NHANES 1999-2000 to 2013-2014. Obesity (Silver Spring). 2017 Apr;25(4):739-746. doi: 10.1002/oby.21782. Epub 2017 Feb 28. PMID 28245098
- [Background] Freedman DS, Butte NF, Taveras EM, Goodman AB, Ogden CL, Blanck HM. The Limitations of Transforming Very High Body Mass Indexes into z-Scores among 8.7 Million 2- to 4-Year-Old Children. J Pediatr. 2017 Sep;188:50-56.e1. doi: 10.1016/j.jpeds.2017.03.039. Epub 2017 Apr 19. PMID 28433203
- [Background] Freedman DS, Butte NF, Taveras EM, Goodman AB, Blanck HM. Longitudinal changes in BMI z-scores among 45 414 2-4-year olds with severe obesity. Ann Hum Biol. 2017 Dec;44(8):687-692. doi: 10.1080/03014460.2017.1388845. Epub 2017 Oct 30. PMID 29082754
- [Background] Freedman DS, Berenson GS. Tracking of BMI z Scores for Severe Obesity. Pediatrics. 2017 Sep;140(3):e20171072. doi: 10.1542/peds.2017-1072. Epub 2017 Aug 22. PMID 28830920
- [Background] Gattshall ML, Shoup JA, Marshall JA, Crane LA, Estabrooks PA. Validation of a survey instrument to assess home environments for physical activity and healthy eating in overweight children. Int J Behav Nutr Phys Act. 2008 Jan 11;5:3. doi: 10.1186/1479-5868-5-3. PMID 18190709
- [Background] Martin-Garcia M, Vila-Maldonado S, Rodriguez-Gomez I, Faya FM, Plaza-Carmona M, Pastor-Vicedo JC, Ara I. The Spanish version of the Three Factor Eating Questionnaire-R21 for children and adolescents (TFEQ-R21C): Psychometric analysis and relationships with body composition and fitness variables. Physiol Behav. 2016 Oct 15;165:350-7. doi: 10.1016/j.physbeh.2016.08.015. Epub 2016 Aug 15. PMID 27538345
- [Background] Cappelleri JC, Bushmakin AG, Gerber RA, Leidy NK, Sexton CC, Lowe MR, Karlsson J. Psychometric analysis of the Three-Factor Eating Questionnaire-R21: results from a large diverse sample of obese and non-obese participants. Int J Obes (Lond). 2009 Jun;33(6):611-20. doi: 10.1038/ijo.2009.74. Epub 2009 Apr 28. PMID 19399021
- [Background] Scott SN, Springer CM, Oody JF, McClanahan MS, Wiseman BD, Kybartas TJ, Coe DP. Development and Validation of a PACER Prediction Equation for VO2peak in 10- to 15-Year-Old Youth. Pediatr Exerc Sci. 2019 May 1;31(2):223-228. doi: 10.1123/pes.2018-0136. Epub 2019 Jan 3. PMID 30606067
- [Background] Welk, G.J. and M.D. Meredith, eds. Fitnessgram / Activitygram Reference Guide. 2008, The Cooper Institute.: Dallas, TX.
- [Background] Blumberg SJ, Bialostosky K, Hamilton WL, Briefel RR. The effectiveness of a short form of the Household Food Security Scale. Am J Public Health. 1999 Aug;89(8):1231-4. doi: 10.2105/ajph.89.8.1231. PMID 10432912
- [Background] Mills SD, Malcarne VL, Fox RS, Sadler GR. Psychometric Evaluation of the Brief Acculturation Scale for Hispanics. Hisp J Behav Sci. 2014 May 1;36(2):164-174. doi: 10.1177/0739986314526697. PMID 25110387
- [Background] Villarreal, R., S. Blozis, and K. Widaman, Factorial Invariance of a Pan-Hispanic Familism Scale. Hispanic Journal of Behavioral Sciences, 2005. 27: p. 409 - 425.
- [Background] Knight GP, Gonzales NA, Saenz DS, Bonds DD, German M, Deardorff J, Roosa MW, Updegraff KA. The Mexican American Cultural Values scales for Adolescents and Adults. J Early Adolesc. 2010 Jun;30(3):444-481. doi: 10.1177/0272431609338178. PMID 20644653
- [Background] Zeller MH, Modi AC. Development and initial validation of an obesity-specific quality-of-life measure for children: sizing me up. Obesity (Silver Spring). 2009 Jun;17(6):1171-7. doi: 10.1038/oby.2009.47. Epub 2009 Mar 5. PMID 19265795
- [Background] Prescott CA, McArdle JJ, Hishinuma ES, Johnson RC, Miyamoto RH, Andrade NN, Edman JL, Makini GK Jr, Nahulu LB, Yuen NY, Carlton BS. Prediction of major depression and dysthymia from CES-D scores among ethnic minority adolescents. J Am Acad Child Adolesc Psychiatry. 1998 May;37(5):495-503. doi: 10.1097/00004583-199805000-00012. PMID 9585651
- [Background] Soler J, Perez-Sola V, Puigdemont D, Perez-Blanco J, Figueres M, Alvarez E. [Validation study of the Center for Epidemiological Studies-Depression of a Spanish population of patients with affective disorders]. Actas Luso Esp Neurol Psiquiatr Cienc Afines. 1997 Jul-Aug;25(4):243-9. Spanish. PMID 9412163
- [Background] Garrison CZ, Addy CL, Jackson KL, McKeown RE, Waller JL. The CES-D as a screen for depression and other psychiatric disorders in adolescents. J Am Acad Child Adolesc Psychiatry. 1991 Jul;30(4):636-41. doi: 10.1097/00004583-199107000-00017. PMID 1890099
- [Background] Faulstich ME, Carey MP, Ruggiero L, Enyart P, Gresham F. Assessment of depression in childhood and adolescence: an evaluation of the Center for Epidemiological Studies Depression Scale for Children (CES-DC). Am J Psychiatry. 1986 Aug;143(8):1024-7. doi: 10.1176/ajp.143.8.1024. PMID 3728717
- [Background] Moyers TB, Rowell LN, Manuel JK, Ernst D, Houck JM. The Motivational Interviewing Treatment Integrity Code (MITI 4): Rationale, Preliminary Reliability and Validity. J Subst Abuse Treat. 2016 Jun;65:36-42. doi: 10.1016/j.jsat.2016.01.001. Epub 2016 Jan 13. PMID 26874558
- [Background] Rabin BA, McCreight M, Battaglia C, Ayele R, Burke RE, Hess PL, Frank JW, Glasgow RE. Systematic, Multimethod Assessment of Adaptations Across Four Diverse Health Systems Interventions. Front Public Health. 2018 Apr 9;6:102. doi: 10.3389/fpubh.2018.00102. eCollection 2018. PMID 29686983
- [Background] Ritzwoller DP, Sukhanova A, Gaglio B, Glasgow RE. Costing behavioral interventions: a practical guide to enhance translation. Ann Behav Med. 2009 Apr;37(2):218-27. doi: 10.1007/s12160-009-9088-5. Epub 2009 Mar 17. PMID 19291342
- [Background] Cidav Z, Mandell D, Pyne J, Beidas R, Curran G, Marcus S. A pragmatic method for costing implementation strategies using time-driven activity-based costing. Implement Sci. 2020 May 5;15(1):28. doi: 10.1186/s13012-020-00993-1. PMID 32370752
- [Background] Mauricio AM, Tein JY, Gonzales NA, Millsap RE, Dumka LE. Attendance Patterns and Links to Non-Response on Child Report of Internalizing among Mexican-Americans Randomized to a Universal Preventive Intervention. Prev Sci. 2018 Feb;19(Suppl 1):27-37. doi: 10.1007/s11121-016-0632-9. PMID 26786469
- [Background] Turer CB, Stroo M, Brouwer RJ, Krause KM, Lovelady CA, Bastian LA, Peterson B, Ostbye T. Do high-risk preschoolers or overweight mothers meet AAP-recommended behavioral goals for reducing obesity? Acad Pediatr. 2013 May-Jun;13(3):243-50. doi: 10.1016/j.acap.2013.01.003. Epub 2013 Jan 9. PMID 23491583
- [Background] Rich SS, DiMarco NM, Huettig C, Essery EV, Andersson E, Sanborn CF. Perceptions of health status and play activities in parents of overweight Hispanic toddlers and preschoolers. Fam Community Health. 2005 Apr-Jun;28(2):130-41. doi: 10.1097/00003727-200504000-00005. PMID 15778627
- [Background] Hernandez RG, Cheng TL, Serwint JR. Parents' healthy weight perceptions and preferences regarding obesity counseling in preschoolers: pediatricians matter. Clin Pediatr (Phila). 2010 Aug;49(8):790-8. doi: 10.1177/0009922810368288. Epub 2010 Jun 3. PMID 20522610
- [Background] Gauthier KI, Gance-Cleveland B. Hispanic parents' perceptions of their preschool children's weight status. J Spec Pediatr Nurs. 2016 Apr;21(2):84-93. doi: 10.1111/jspn.12143. Epub 2016 Apr 15. PMID 27079822
- [Background] McGavock J, Chauhan BF, Rabbani R, Dias S, Klaprat N, Boissoneault S, Lys J, Wierzbowski AK, Sakib MN, Zarychanski R, Abou-Setta AM. Layperson-Led vs Professional-Led Behavioral Interventions for Weight Loss in Pediatric Obesity: A Systematic Review and Meta-analysis. JAMA Netw Open. 2020 Jul 1;3(7):e2010364. doi: 10.1001/jamanetworkopen.2020.10364. PMID 32658289
- [Background] Bleich SN, Segal J, Wu Y, Wilson R, Wang Y. Systematic review of community-based childhood obesity prevention studies. Pediatrics. 2013 Jul;132(1):e201-10. doi: 10.1542/peds.2013-0886. Epub 2013 Jun 10. PMID 23753099
- [Background] Haemer, M., Why Does Cooking Matter? Outcomes of Nutrition Education in Collaboration with Health Care, in Share Our Strength's National Convening. 2015: Washington DC.
- [Background] Li PP, Mackey G, Callender C, Dave JM, Olvera N, Alford S, Thompson D. Culinary Education Programs for Children in Low-Income Households: A Scoping Review. Children (Basel). 2020 May 13;7(5):47. doi: 10.3390/children7050047. PMID 32414003
- [Background] Hasan B, Thompson WG, Almasri J, Wang Z, Lakis S, Prokop LJ, Hensrud DD, Frie KS, Wirtz MJ, Murad AL, Ewoldt JS, Murad MH. The effect of culinary interventions (cooking classes) on dietary intake and behavioral change: a systematic review and evidence map. BMC Nutr. 2019 May 10;5:29. doi: 10.1186/s40795-019-0293-8. eCollection 2019. PMID 32153942
- [Background] Overcash F, Ritter A, Mann T, Mykerezi E, Redden J, Rendahl A, Vickers Z, Reicks M. Impacts of a Vegetable Cooking Skills Program Among Low-Income Parents and Children. J Nutr Educ Behav. 2018 Sep;50(8):795-802. doi: 10.1016/j.jneb.2017.10.016. Epub 2017 Dec 12. PMID 29242140
- [Background] Liu GC, Hannon T, Qi R, Downs SM, Marrero DG. The obesity epidemic in children: Latino children are disproportionately affected at younger ages. Int J Pediatr Adolesc Med. 2015 Mar;2(1):12-18. doi: 10.1016/j.ijpam.2015.03.004. Epub 2015 Apr 4. PMID 30805430
- [Background] Lee H, Hicken MT. Cumulative social risk and racial/ethnic disparities in obesity during the transition to adulthood. J Health Care Poor Underserved. 2013 May;24(2):907-27. doi: 10.1353/hpu.2013.0090. PMID 23728056
- [Background] Dabelea D, Mayer-Davis EJ, Saydah S, Imperatore G, Linder B, Divers J, Bell R, Badaru A, Talton JW, Crume T, Liese AD, Merchant AT, Lawrence JM, Reynolds K, Dolan L, Liu LL, Hamman RF; SEARCH for Diabetes in Youth Study. Prevalence of type 1 and type 2 diabetes among children and adolescents from 2001 to 2009. JAMA. 2014 May 7;311(17):1778-86. doi: 10.1001/jama.2014.3201. PMID 24794371
- [Background] Maskarinec G, Grandinetti A, Matsuura G, Sharma S, Mau M, Henderson BE, Kolonel LN. Diabetes prevalence and body mass index differ by ethnicity: the Multiethnic Cohort. Ethn Dis. 2009 Winter;19(1):49-55. PMID 19341163
- [Background] Aguayo-Mazzucato C, Diaque P, Hernandez S, Rosas S, Kostic A, Caballero AE. Understanding the growing epidemic of type 2 diabetes in the Hispanic population living in the United States. Diabetes Metab Res Rev. 2019 Feb;35(2):e3097. doi: 10.1002/dmrr.3097. Epub 2018 Dec 4. PMID 30445663
- [Background] O'Connor EA, Evans CV, Burda BU, Walsh ES, Eder M, Lozano P. Screening for Obesity and Intervention for Weight Management in Children and Adolescents: Evidence Report and Systematic Review for the US Preventive Services Task Force. JAMA. 2017 Jun 20;317(23):2427-2444. doi: 10.1001/jama.2017.0332. PMID 28632873
- [Background] Weaver RG, Brazendale K, Hunt E, Sarzynski MA, Beets MW, White K. Disparities in childhood overweight and obesity by income in the United States: an epidemiological examination using three nationally representative datasets. Int J Obes (Lond). 2019 Jun;43(6):1210-1222. doi: 10.1038/s41366-019-0331-2. Epub 2019 Feb 4. PMID 30718822
- [Background] Kelly ML, Ackerman PD, Ross LF. The participation of minorities in published pediatric research. J Natl Med Assoc. 2005 Jun;97(6):777-83. PMID 16035575
- [Background] Love-Osborne K, Fortune R, Sheeder J, Federico S, Haemer MA. School-based health center-based treatment for obese adolescents: feasibility and body mass index effects. Child Obes. 2014 Oct;10(5):424-31. doi: 10.1089/chi.2013.0165. Epub 2014 Sep 26. PMID 25259781
- [Background] Fagg J, Chadwick P, Cole TJ, Cummins S, Goldstein H, Lewis H, Morris S, Radley D, Sacher P, Law C. From trial to population: a study of a family-based community intervention for childhood overweight implemented at scale. Int J Obes (Lond). 2014 Oct;38(10):1343-9. doi: 10.1038/ijo.2014.103. Epub 2014 Jun 12. PMID 24919564
- [Background] Sacher PM, Kolotourou M, Chadwick PM, Cole TJ, Lawson MS, Lucas A, Singhal A. Randomized controlled trial of the MEND program: a family-based community intervention for childhood obesity. Obesity (Silver Spring). 2010 Feb;18 Suppl 1:S62-8. doi: 10.1038/oby.2009.433. PMID 20107463
- [Background] Hoelscher DM, Butte NF, Barlow S, Vandewater EA, Sharma SV, Huang T, Finkelstein E, Pont S, Sacher P, Byrd-Williams C, Oluyomi AO, Durand C, Li L, Kelder SH. Incorporating primary and secondary prevention approaches to address childhood obesity prevention and treatment in a low-income, ethnically diverse population: study design and demographic data from the Texas Childhood Obesity Research Demonstration (TX CORD) study. Child Obes. 2015 Feb;11(1):71-91. doi: 10.1089/chi.2014.0084. Epub 2015 Jan 2. PMID 25555188
- [Background] Butte NF, Hoelscher DM, Barlow SE, Pont S, Durand C, Vandewater EA, Liu Y, Adolph AL, Perez A, Wilson TA, Gonzalez A, Puyau MR, Sharma SV, Byrd-Williams C, Oluyomi A, Huang T, Finkelstein EA, Sacher PM, Kelder SH. Efficacy of a Community- Versus Primary Care-Centered Program for Childhood Obesity: TX CORD RCT. Obesity (Silver Spring). 2017 Sep;25(9):1584-1593. doi: 10.1002/oby.21929. Epub 2017 Jul 13. PMID 28703504
- [Background] Chambers DA. Sharpening our focus on designing for dissemination: Lessons from the SPRINT program and potential next steps for the field. Transl Behav Med. 2020 Dec 31;10(6):1416-1418. doi: 10.1093/tbm/ibz102. PMID 31313812
- [Background] Hollingworth W, Hawkins J, Lawlor DA, Brown M, Marsh T, Kipping RR. Economic evaluation of lifestyle interventions to treat overweight or obesity in children. Int J Obes (Lond). 2012 Apr;36(4):559-66. doi: 10.1038/ijo.2011.272. Epub 2012 Jan 17. PMID 22249222
- [Background] Polgar, J., S. Goldberg, and M. Haemer, An Economic Perspective On a Community-Based Childhood Obesity Treatment Program, in Colorado Public Health Forum. 2016: Aurora, CO
- [Background] Haemer MA, Ranade D, Baron AE, Krebs NF. A clinical model of obesity treatment is more effective in preschoolers and Spanish speaking families. Obesity (Silver Spring). 2013 May;21(5):1004-12. doi: 10.1002/oby.20192. PMID 23784904
- [Background] S, A., et al., Boot Camp Translation for the Prevention of Type 2 Diabetes (T2D) in Fort Collins' Hispanic/Latino Adolescents., in CCTSI Community Engagement Conference. 2017
- [Background] Haemer, M., et al., Pilot Results of a Multi-level Partnership to treat Obesity in Low-Income Hispanic Children, in The Obesity Society Annual Meeting. 2011. p. publication # LB-P-50
- [Background] Haemer, M., et al. An Enhanced Screen Performs Better than 5-2-1-0 for Lifestyle Assessment in Low-Income Hispanic Children. in Pediatric Academic Societies. 2012. Boston, MA
- [Background] Haemer, M., et al. One-Year Outcomes from a Controlled Trial of Family-Inclusive Weight Management in Underserved Children. in Pediatric Academic Societies. 2015. San Diego, CA
- [Background] Haemer, M., et al., Food Neophobia in Latino Preschoolers: Correlation with Intake and Pilot Intervention Results, in American Society of Nutrition Annual Meeting at Experimental Biology. 2014: San Diego, CA
- [Background] Belay B, Frintner MP, Liebhart JL, Lindros J, Harrison M, Sisk B, Dooyema CA, Hassink SG, Cook SR. US Pediatrician Practices and Attitudes Concerning Childhood Obesity: 2006 and 2017. J Pediatr. 2019 Aug;211:78-84.e2. doi: 10.1016/j.jpeds.2019.04.030. Epub 2019 May 18. PMID 31113716
- [Background] Welk GJ, Meredith MD, Ihmels M, Seeger C. Distribution of health-related physical fitness in Texas youth: a demographic and geographic analysis. Res Q Exerc Sport. 2010 Sep;81(3 Suppl):S6-15. doi: 10.1080/02701367.2010.10599689. PMID 21049833
- [Derived] Haemer M, Tong S, Bracamontes P, Gritz M, Osborn B, Perez-Jolles M, Shomaker L, Steen E, Studts C, Boles R. Randomized-controlled trial of a whole-family obesity prevention and treatment intervention designed for low-income Hispanic families: HeLP the healthy living program. Contemp Clin Trials. 2023 Dec;135:107359. doi: 10.1016/j.cct.2023.107359. Epub 2023 Oct 16. PMID 37852530
- See also: Evidence Synthesis, No. 150: Screening for Obesity and Interventions for Weight Management in Children and Adolescents: A Systematic Evidence Review for the U.S. Preventive Services Task Force : Agency for Healthcare Research and Quality (US) — http://www.ncbi.nlm.nih.gov/books/NBK476325/
- See also: USDA. Food Security in the U.S. - Survey Tools. — https://www.ers.usda.gov/topics/food-nutrition-assistance/food-security-in-the-us/survey-tools/
- See also: FITNESSGRAM by GreenLight Fitness — https://www.fitnessgram.net/
- See also: Pew Research Center - Hispanic Trends. Demographic and Economic Profiles of Hispanics by State and County, 2014. 2020 — http://www.pewresearch.org/hispanic/states/state/co
- See also: Share_our_Strength. Cooking Matters Hands-On Cooking Courses. [web page] 2019 — http://cookingmatters.org
- See also: US_Census_Bureau. Detailed Languages Spoken at Home and Ability to Speak English for the Population 5 Years and Over: 2009-2013. 2015 Oct 28, 2015 — https://data.census.gov/cedsci/table?q=Language%20Spoken%20at%20Home&tid=ACSST1Y2019.S1601&hidePreview=true
- See also: ServSafe. ServSafe - Food Safety Training. 2020 2020 — https://www.servsafe.com/ServSafe-Food-Handler/Buy-Handler-Products?gclid=Cj0KCQjwy8f6BRC7ARIsAPIXOjj0S3lIjS62X_ltKs9nyPRBUSZ_RofVDOdJtz3POiNCU0YRcThiIqcaAlcVEALw_wcB

DOCUMENTS (3):
  • Informed Consent Form: Consent-Parents (2021-07-16): https://cdn.clinicaltrials.gov/large-docs/55/NCT05041855/ICF_000.pdf
  • Informed Consent Form: Consent-HeLP Staff (2021-07-16): https://cdn.clinicaltrials.gov/large-docs/55/NCT05041855/ICF_001.pdf
  • Informed Consent Form: Consent-Providers (2021-07-16): https://cdn.clinicaltrials.gov/large-docs/55/NCT05041855/ICF_002.pdf